CLINICAL TRIAL: NCT02744066
Title: A Pilot Study to Evaluate Patient Tolerance and Nursing Ease-of-Use of a Novel Hearing Protection Device to Reduce Exposure to Excessive Noise Among Patients Undergoing Neonatal Intensive Care
Brief Title: A Pilot Study to Evaluate Patient Tolerance and Nursing Ease-of-Use of a Novel Hearing Protection Device
Acronym: NEATCAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Balsan, MD (Other)
Responsible Party: Sponsor-Investigator, Michael Balsan, MD, Associate Professor of Pediatrics, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PRO16010220
Record Dates: First submitted 2016-04-14; First posted 2016-04-20 (Estimated); Results first posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Hearing Impairment
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Neonates (Other): Neonates admitted to the NICU will be fitted for NEATCAP, non-invasive novel hearing protection device.
  Interventions: Device: NEATCAP

INTERVENTIONS:
Device: NEATCAP — Neonates will be sized and fitted to wear the non-invasive novel hearing protection device over a set period of time in the NICU. Vitals will be monitored.

SUMMARY:
Before they are born, babies are protected from hearing very loud noises by their mother's bodies. After delivery, they are exposed to many loud noises that are potentially harmful. These noises happen in the neonatal intensive care unit (NICU). The purpose of this research project is to test the fit and the ease-of-use of a new device that may protect infant's hearing in the NICU.

DETAILED DESCRIPTION:
Despite the best efforts of Neonatal Intensive Care Unit (NICU) caregivers, vulnerable and fragile NICU patients are frequently exposed to noxious levels of noise from monitoring and respiratory equipment alarms, as well as from routine NICU care practices. Particularly detrimental to sleep and auditory development are patient exposures to high frequency noises that are specifically designed to alert NICU caregivers to important changes in patient status. This pilot study will help evaluate the fit, ergonomic design and the ease-of-use of a novel hearing protection system (special ear-muffs along with a unique attachment mechanism) specifically designed top diminish the transmission of high frequency noises to patients within the NICU, while allowing some transmission of low frequency sounds, such as a mother's voice.

ELIGIBILITY:
Inclusion Criteria:

* Neonate admitted to the Neonatal Intensive Care Unit
* Age greater than 12 hours and less than 2 weeks
* Informed consent from the parent(s)

Exclusion Criteria:

* Significant cranial trauma noted on admission
* Congenital anomalies of the head and/or neck
* Hemodynamic instability requiring pharmacologic intervention
* Recommendation by the attending neonatologist not to enroll the patient

Ages: 12 Hours to 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2017-10-05 (Actual); Study Completion 2017-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Balsan, MD, Principal Investigator — Principal Investigator
Locations (1):
- Magee Womens, UPMC Hamot, Erie, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Balsan MJ, Burns J, Kimock F, Hirsch E, Unger A, Telesco R, Bloch-Salisbury E. A pilot study to assess the safety, efficacy and ease of use of a novel hearing protection device for hospitalized neonates. Early Hum Dev. 2021 May;156:105365. doi: 10.1016/j.earlhumdev.2021.105365. Epub 2021 Mar 26. PMID 33857731

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from admissions to the neonatal intensive care unit (NICU) in two phases. In phase #1 of the study 25 infants were recruited for participation and 25 infants completed the protocol. In phase #2 of the study 30 additional infants were recruited, with 25 infants completing the protocol. The total number studied was 50.
Groups:
- Phase #1: Infants recruited in phase #1 had the device placed for 1 hour, with recordings of vital signs before and after devise placement.
- Phase #2: Infants recruited in phase #2 had the device placed for 8 hour periods on three consecutive days with vital signs recorded before, during and after device placements.
Period: Overall Study
Arm/Group | Phase #1 | Phase #2
Started | 25 | 30
Completed | 25 | 25
Not Completed | 0 | 5
Not completed — Withdrawal by parent | 0 | 1
Not completed — Discharged from NICU prior to completion | 0 | 4

BASELINE CHARACTERISTICS:
Population: 25 patients recruited for the study for phase #1 and 25 patient outcomes analyzed for phase #1. 30 additional patients recruited for the study in phase #2 and 25 patient outcomes analyzed for phase #2.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase #1 | Phase #2 | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25 | 25 | 50
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 15 | 17 | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Gestational Age at Birth [Mean (Standard Deviation); unit: Weeks] — Mean gestational age at birth in weeks
  Weeks | 36.6 (3.29) | 34.8 (3.87) | 35.7 (3.7)
Birth Weight [Mean (Standard Deviation); unit: kilograms] — Birth Weight in kilograms
  kilograms | 2.6 (0.84) | 2.3 (0.94) | 2.5 (0.9)
Head Circumference [Mean (Standard Deviation); unit: centimeters] — Occipital-Frontal Head Circumference at birth
  centimeters | 32.3 (3.03) | 31.4 (3.66) | 31.8 (3.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Skin Erythema After Device Application
Description: Skin will be assessed for adverse effects such as any device-related adverse events, including evidence of skin redness, rash and/or bruising or discomfort at the site of device application. Skin erythema was described as none, mild, moderate or severe as evaluated by the NICU nursing staff.
Time Frame: Skin erythema was evaluated at the time of device removal after 1 hour of application in phase #1 and after 3 daily 8 hour periods of application in phase #2.
Population: Phase #2 data reports the number of participants experiencing erythema at any time after device removal after 3 daily 8 hour periods of device application.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase #1 | Phase #2
Number analyzed (Participants) | 25 | 25
Participants
  Skin Erythema after Device Application: No Skin Erythema | 10 | 10
  Skin Erythema after Device Application: Mild Skin Erythema | 15 | 14
  Skin Erythema after Device Application: Moderate Skin Erythema | 0 | 0
  Skin Erythema after Device Application: Severe Skin Erythema | 0 | 1
  Skin Erythema after Device Application: Skin Breakdown | 0 | 0
  Skin Erythema at Baseline: No Skin Erythema | 25 | 25
  Skin Erythema at Baseline: Mild Skin Erythema | 0 | 0
  Skin Erythema at Baseline: Moderate Skin Erythema | 0 | 0
  Skin Erythema at Baseline: Severe Skin Erythema | 0 | 0
  Skin Erythema at Baseline: Skin Breakdown | 0 | 0

2. Secondary Outcome: Number of Participants With Specific Responses to the Ease of Use Questionnaire for NICU Staff.
Description: A >80% positive response to a multi-question Ease-of-Use Questionnaire completed by the participating NICU staff. Ease-of-Use Questionnaire constructed on a 5 point Likert Scale: 1 = Strongly Disagree, 2 = Disagree, 3 = Neutral, 4 = Agree, 5 = Strongly Agree that the device was easy-to-use. Phase #1 consists of 25 data points. Phase #2 consists of 25 data points. Evaluations were obtained after device removal in both phases.
Time Frame: After 1 hour in phase #1 / After 3 x 8 hours in phase #2
Measure: Count of Participants; unit: Participants
Groups:
- Phase #1: Infants recruited in phase #1 had the device placed for 1 hour.
- Phase #2: Infants recruited in phase #2 had the device placed daily for the same 8 hour periods on three consecutive days.
Arm/Group | Phase #1 | Phase #2
Number analyzed (Participants) | 25 | 25
Participants
  Strongly Disagree | 0 | 0
  Disagree | 0 | 0
  Neutral | 0 | 1
  Agree | 4 | 10
  Strongly Agree | 21 | 14

ADVERSE EVENTS:
Time Frame: Adverse event data were collected immediately after device removal for both arms of the study.
Description: Systematic Assessment of the skin condition of study subjects by participating NICU nurses was conducted per protocol for 25 infants in phase #1 and 25 infants in phase #2.
Arm/Group | Phase #1 | Phase #2
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 1/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase #1 (N=25) | Phase #2 (N=25)
Severe Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Significant but transient erythema associated with device placement without evidence of skin breakdown

LIMITATIONS AND CAVEATS:
Limited number of very low birth weight infants in the available study population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-28): https://cdn.clinicaltrials.gov/large-docs/66/NCT02744066/Prot_SAP_000.pdf